CLINICAL TRIAL: NCT01692132
Title: A Study on the Safety and Effectiveness of Prucalopride in the Treatment of Chronic Constipation
Brief Title: A Post Marketing Surveillance Study on the Safety and Effectiveness of Prucalopride in the Treatment of Chronic Constipation
Status: Withdrawn | Type: Observational
Why Stopped: The company decided to cancel this study in conformity with PH FDA Circular 2013-004
Sponsor: Janssen Pharmaceutica (Industry)
Responsible Party: Sponsor
Other Study IDs: CR017521; PRUCOP4001 (Other: Janssen Pharmaceutica)
Record Dates: First submitted 2012-09-20; First posted 2012-09-25 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Constipation
Keywords: Chronic Constipation; Prucalopride; Post Marketing Surveillance
MeSH Terms: interventions — prucalopride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prucalopride
  Interventions: Drug: Prucalopride

INTERVENTIONS:
Drug: Prucalopride — Prucalopride 2 mg tablet/day orally for 12 weeks. For elderly patients (>65 years old), patients with renal impairment not requiring dialysis or patients with severe hepatic impairment, 1mg prucalopride once daily should be given.

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of prucalopride in the treatment of Filipino patients with chronic constipation whom prior laxatives fail to provide adequate relief.

DETAILED DESCRIPTION:
This is a 12-week open label (all people know the identity of the intervention), multi-center, prospective (the patients are identified and then followed forward in time for the outcome of the study) observational study assessing the safety and effectiveness of prucalopride among Filipino patients with chronic constipation. Chronic constipation is a condition in which bowel movements are infrequent or incomplete for a prolonged time. The use of prucalopride should be used in accordance with the approved product label and will follow the normal medical practice of the investigators. Patients should take 2 mg prucalopride tablet orally once daily. For elderly patients (>65 years old), patients with renal impairment not requiring dialysis or patients with severe hepatic impairment, 1mg prucalopride once daily should be given. Patients will be asked to fill-up a patient diary daily for 12-weeks to monitor the bowel movement during the study period. All adverse events and concomitant medications taken by the patients during the study will be documented accordingly. Patients will be monitored during the 12-week period of observation while the patients are in prucalopride treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic constipation by history and physical examination, including rectal exam
* History of chronic constipation not satisfied with laxatives
* Patient reports, on average, 2 or fewer spontaneous bowel movements (SBMs) per week and 1 or more of the following for the last three months: very hard (little balls) and/or hard stools in more than 25% of bowel movements (BMs); sensation of incomplete evacuation in more than 25% of BMs; straining at defecation in more than 25% of BMs; sensation of ano-rectal obstruction or blockade in more than 25% of BMs; a need for digital manipulation to facilitate evacuation in more than 25% of BMs
* Females of childbearing potential agree to use highly effective contraceptive methods

Exclusion Criteria:

* Renal impairment requiring dialysis
* Secondary chronic constipation and organic gastrointestinal (GI) disorders
* Intestinal perforation / obstruction due to structural or functional disorder of the gut wall, obstructive ileus, severe inflammatory condition of the intestinal tract such as Crohn's disease, ulcerative colitis, toxic megacolon / rectum
* Hypersensitive to Prucalopride or to any of its components
* Patients receiving concomitant drugs known to cause QTc prolongation
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Filipino patients with chronic constipation
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-02; Primary Completion 2014-02 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of patients discontinuing treatment due to adverse events, serious adverse events, or adverse drug reactions | 12 weeks

SECONDARY OUTCOMES:
The percentage of patients having at least 3 spontaneous complete bowel movements (SCBM) in a week after treatment with prucalopride | 12 weeks
  SCBM is defined as a sense of complete evacuation of bowel without straining.
The change from baseline in the Patient Assessment of Constipation Symptoms (PAC-SYM) score after treatment with prucalopride | Baseline, 12 weeks
  The PAC-SYM questionnaire is a 12-item survey that measures constipation symptoms and associated severity across three domains: stool symptoms, rectal symptoms, and abdominal symptoms. Symptom items are rated on a 5-point Likert severity scale. Item values are scored from 0 to 4, with 0 indicating absence of symptom, 1 = mild, 2 = moderate, 3 = severe, and 4 = very severe indicating the worst severity of that symptom.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica Clinical Trial, Study Director — Janssen Pharmaceutica
Locations (7):
- Philippines (7):
  - City of Muntinlupa
  - City of Taguig
  - Makati City
  - Manila
  - Marikina City
  - Quezon City
  - San Juan City